CLINICAL TRIAL: NCT02940093
Title: Implementation of a Pipeline Integrating Gut Metagenome Data, Host Immunogenetic Characteristics and Clinical Gut Inflammatory Biomarkers for Stratified Clinical Management
Brief Title: Pipeline Integrating Gut Metagenome Data, Host Immunogenetic Characteristics and Clinical Gut Inflammatory Biomarkers
Acronym: ImMiGeNe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: ImMiGeNe-001
Record Dates: First submitted 2016-10-13; First posted 2016-10-20 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Stem Cell Transplantation
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Feces Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Stem cell transplant recipient
  Interventions: Other: Stem cell transplantation
- Stem cell donor

INTERVENTIONS:
Other: Stem cell transplantation — Intervention is not conducted as part of the study but patients at Tübingen University Hospital undergoing this intervention as part of their standard care are being monitored in this observational study.
  Groups: Stem cell transplant recipient

SUMMARY:
The combined analysis of microbiome, immunological parameters and host genetics in patients has potential for applying personalized approaches of prevention, diagnostics or therapy in the future. However, the acquisition and analysis of these patient characteristics in a scientifically sound, technically reliable, cost-effective, practicable and future-oriented fashion are a far from trivial task. Therefore the objectives of the study are (i) to optimize a sample and data acquisition and analysis pipeline that fulfills these criteria (using samples from healthy volunteers); (ii) validate the pipeline in a cohort of children undergoing stem cell transplantation, yielding information on host immuno-genetics, gut immune function and the human gut microbiome; (iii) deduct the most critical parameters for host-microbiome interplay from this complex dataset.

ELIGIBILITY:
Inclusion Criteria:

* Patient (stem cell recipient) with hematological malignancies, age 3-18
* Healthy allogeneic stem cell donor (identical or non-identical related donor)

Exclusion Criteria:

* Patients <3 years of age
* Patient who are unable to provide urine, stool or blood samples due to their medical condition

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients undergoing stem cell transplantation due to hematological malignancies Allogeneic stem cell donors
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11-24 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Immune system - intestinal microbiota co-re-emergence after myeloablative conditioning and antibiotics treatment, respectively. | through study completion, anticipated after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander NR Weber, PhD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Children's Hospital Tübingen, Tübingen, Germany